CLINICAL TRIAL: NCT03746795
Title: Realization of Spirometry Measurement Using Electrical Impedance Tomography (EIT)
Brief Title: Spirometry Using Electrical Impedance Tomography
Acronym: EIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EITspiro
Record Dates: First submitted 2018-11-13; First posted 2018-11-20 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: electrical impedance tomography; spirometric examination; bioimpedance; FVC; FEV1; Tiffeneau index

STUDY DESIGN:
Intervention Model Description: During the experiment, six measurements will be performed for each examined individual to calculate the spirometric parameters of FVC, FEV1 and Tiffenea's index (TI) FEV1/FVC. Spirometry measurements will be performed in a randomized order: two standard spirometric examinations, two spirometric examinations using EIT and two simultaneous measurements using both methods.
  Each subject will undergo all six measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard spirometry (No Intervention): Standard spirometry measurement with a pneumotachograph alone.
- EIT alone (Experimental): Spirometric examinations realized using the EIT
  Interventions: Device: Spirometric examinations realized using the EIT
- Simultaneous standard spirometry and EIT (Experimental): Simultaneous measurement by spirometer and EIT
  Interventions: Device: Simultaneous measurement by spirometer and EIT

INTERVENTIONS:
Device: Spirometric examinations realized using the EIT — Spirometric examinations will be realized using the EIT alone.
  Arms: EIT alone
Device: Simultaneous measurement by spirometer and EIT — Spirometric examinations will be realized using the simultaneous measurement by spirometer and EIT
  Arms: Simultaneous standard spirometry and EIT

SUMMARY:
The main aim of this study is to test spirometry measurements using EIT with a calibration using tidal volume obtained from the simultaneous standard spirometry measurement. Another goal is to compare, based on the calibration, the spirometry parameters obtained from separate measurements using EIT and the standard spirometry using a pneumotachograph.

All spirometry measurements will be conducted in accordance with the latest available standards of the American Thoracic Society (ATS) and European Respiratory Society (ERS) from the year 2005, including their emendation from 2017.

DETAILED DESCRIPTION:
Adding the pneumotachograph and antibacterial filter to the respiratory system can lead to increased dead space, flow resistance, and change the respiratory pattern. All of these negative features and reduced patient co-operation affect the measured results and their interpretation. The aim of this study is to test spirometry measurement using EIT and evaluate such spirometry parameters as forced vital capacity (FVC), forced expiratory volume exhaled in the first second of a forced expiration (FEV1) and ratio of FEV1/FVC called Tiffeneau index (TI) based on recalculation using the calibration constant. The study will be conducted using Ergostik (Geratherm, Germany) spirometer and EIT system Pulmovista 500 (Dräger, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females > 18 years old
* Signed informed consent has been obtained

Exclusion Criteria:

* Pregnancy
* Cardiac pacemakers
* Electrically active implant
* Critical illness
* Intrathoracic metal implants
* Value of body mass index (BMI)>50

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
FVC | through study completion, an average of 1 year
  forced vital capacity (L)
FEV1 | through study completion, an average of 1 year
  forced expiratory volume exhaled in the first second of a forced expiration (L)
TI | through study completion, an average of 1 year
  ratio of FEV1/FVC called Tiffeneau index (-)

CONTACTS AND LOCATIONS:
Overall Officials: Karel Roubík, prof., Principal Investigator — Czech Technical University in Prague, FBMI
Locations (1):
- Department of Biomedical Technology Faculty of Biomedical Engineering Czech Technical University in Prague, Kladno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
EIT anonymous images and corresponding spirometry data.

REFERENCES:
- [Background] Ngo C, Leonhardt S, Zhang T, Luken M, Misgeld B, Vollmer T, Tenbrock K, Lehmann S. Linearity of electrical impedance tomography during maximum effort breathing and forced expiration maneuvers. Physiol Meas. 2017 Jan;38(1):77-86. doi: 10.1088/1361-6579/38/1/77. Epub 2016 Dec 22. PMID 28004642
- [Background] Vogt B, Lohr S, Zhao Z, Falkenberg C, Ankermann T, Weiler N, Frerichs I. Regional lung function testing in children using electrical impedance tomography. Pediatr Pulmonol. 2018 Mar;53(3):293-301. doi: 10.1002/ppul.23912. Epub 2017 Nov 14. PMID 29136345
- [Background] Lehmann S, Leonhardt S, Ngo C, Bergmann L, Ayed I, Schrading S, Tenbrock K. Global and regional lung function in cystic fibrosis measured by electrical impedance tomography. Pediatr Pulmonol. 2016 Nov;51(11):1191-1199. doi: 10.1002/ppul.23444. Epub 2016 Apr 29. PMID 27127915
- [Background] Vogt B, Zhao Z, Zabel P, Weiler N, Frerichs I. Regional lung response to bronchodilator reversibility testing determined by electrical impedance tomography in chronic obstructive pulmonary disease. Am J Physiol Lung Cell Mol Physiol. 2016 Jul 1;311(1):L8-L19. doi: 10.1152/ajplung.00463.2015. Epub 2016 May 17. PMID 27190067